CLINICAL TRIAL: NCT02514733
Title: Association of Donor Age With Recipient Outcomes in Kidney Transplant
Status: Terminated | Type: Observational
Why Stopped: Due to a lack of laboratory resources, the study was abandoned.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Lorenzo Gallon, Professor in Medicine-Nephrology and Surgery-Organ Transplantation, Northwestern University
Other Study IDs: STU00200153
Record Dates: First submitted 2015-07-28; First posted 2015-08-04 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Complication of Transplant
Keywords: kidney; transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Young donor: Kidney transplant recipient > 60 years of age who received organ from donor <=40 years of age
- Old donor: Kidney transplant recipient >= 60 years of age who received organ from donor >=50 years of age

SUMMARY:
This is a single center study that seeks to study the impact of donor age on recipient outcomes in older kidney transplant recipients.

DETAILED DESCRIPTION:
Over the years use of older kidney allografts has increased in an attempt to bridge the gap between demand and supply of organs. Simultaneously there has been in increase in the number of elderly renal transplant recipients. Numerous factors, both graft and host related, can impact recipient outcomes. The aim of this study is to evaluate the impact of donor age on recipient outcomes, based on the hypothesis is that elderly recipients who receive an older allograft have poorer outcomes that those who receive a younger allograft.

Study subjects will be recruited from the cohort of patients who received a kidney transplant at Northwestern Memorial Hospital.

The transplant clinical database and electronic medical record (OTTR) used in the Comprehensive Transplant Center at Northwestern University will be scanned to screen for kidney transplant recipients who fit the inclusion and exclusion criteria. Potential subjects will then be consented to participate in the study (see attached consent form), and subject participation will be documented in OTTR.

The sample size for the study is 80 subjects, who will be divided into 2 groups based on recipient and donor age. All demographic and clinical data will be collected for the donor and recipients at time of transplant. Follow up clinical data, including but not limited to recipient survival and graft failure will be collected and analyzed for the recipients. Subject confidentiality will be strictly maintained. All subject data will be stored on a secure server and only shared between members of the research team. The investigators plan to publish the results in a peer reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* All adult kidney transplant recipients
* Recipient age > 60 years at the time of transplant
* Transplant was done between January 1, 2013 and December 31, 2014

Exclusion Criteria:

* Recipients of more than one kidney transplant
* Recipients of multi-organ transplants

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All older kidney transplant recipients, age >=60 at transplant who underwent the procedure at Northwestern University during specified time frame ( see below)
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Graft failure | 2 years post transplant
  Graft failure in this study is defined as need for chronic dialysis or re-transplant.

SECONDARY OUTCOMES:
Recipient survival | 2 years post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Gallon, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Comprehensive Transplant Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Knoll GA. Kidney transplantation in the older adult. Am J Kidney Dis. 2013 May;61(5):790-7. doi: 10.1053/j.ajkd.2012.08.049. Epub 2012 Dec 20. PMID 23261121